CLINICAL TRIAL: NCT00003190
Title: Phase III Study of MDR Modulation With PSC-833 (NSC #648265) Followed by Immunotherapy With rIL-2 (NSC #373364) vs. No Further Therapy in Previously Untreated Patients With AML >60 Years
Brief Title: Combination Chemotherapy With or Without Valspodar in Treating Patients With Previously Untreated Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02793; CALGB-9720; U10CA031946 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-10-28 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Cytarabine; Daunorubicin; Etoposide; valspodar

ARMS (2):
- Arm I (cytarabine, daunorubicin, etoposide) (Experimental): Patients receive cytarabine IV continuously over 7 days and daunorubicin IV bolus followed by etoposide IV over 2 hours on days 1-3.
  Interventions: Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: etoposide
- Arm II (valspodar, daunorubicin, etoposide, cytarabine) (Experimental): Patients receive treatment as in arm I with the addition of PSC 833 induction. A loading dose of PSC 833 IV is given over 2 hours, followed by a 74-hour continuous infusion of PSC 833 beginning 2 hours before daunorubicin and etoposide. Patients may receive a second induction course if residual leukemia is present in the bone marrow. Patients who experience a CR and meet certain other criteria receive postremission chemotherapy consisting of cytarabine IV continuously over 5 days plus daunorubicin IV followed by etoposide IV over 2 hours on days 1 and 2. Patients who are randomized to receive PSC 833 during induction chemotherapy receive a loading dose of PSC 833 before beginning a 48-hour continuous infusion of PSC 833 concurrently with cytarabine/daunorubicin/etoposide postremission chemotherapy.
  After completing postremission chemotherapy, patients are randomized to a no further treatment group or IL-2 immunotherapy.
  Interventions: Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: etoposide; Drug: valspodar

INTERVENTIONS:
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: daunorubicin hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; daunomycin hydrochloride; daunorubicin; RP-13057
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: valspodar — Given IV
  Other Names: Amdray; PSC 833
  Arms: Arm II (valspodar, daunorubicin, etoposide, cytarabine)

SUMMARY:
Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without PSC 833 followed by interleukin-2 or no further therapy in treating older patients who have acute myeloid leukemia. Some cancers become resistant to chemotherapy drugs. Combining PSC 833 with more than one chemotherapy drug may reduce resistance to the drugs and allow the cancer cells to be killed. Combining interleukin-2 with combination chemotherapy plus PSC 833 may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the addition of PSC-833 to induction chemotherapy improves complete response rates and whether the addition of PSC-833 to induction and consolidation chemotherapy improves survival for patients with AML >= 60 years.

II. To determine whether the administration of low-dose, subcutaneous rIL-2 immunotherapy with intermittent high-dose boluses after chemotherapy prolongs disease-free survival.

OUTLINE: This is a partially randomized, multicenter study. Patients are stratified according to participating center and disease characteristics (de novo acute myeloid leukemia (AML) versus AML with antecedent myelodysplasia). Patients are randomized to one of two maintenance therapy arms.

Arm I: Patients receive cytarabine IV continuously over 7 days and daunorubicin IV bolus followed by etoposide IV over 2 hours on days 1-3.

Arm II: Patients receive treatment as in arm I with the addition of PSC 833 induction. A loading dose of PSC 833 IV is given over 2 hours, followed by a 74-hour continuous infusion of PSC 833 beginning 2 hours before daunorubicin and etoposide. Patients may receive a second induction course if residual leukemia is present in the bone marrow. Patients who experience a complete remission (CR) and meet certain other criteria receive postremission chemotherapy consisting of cytarabine IV continuously over 5 days plus daunorubicin IV followed by etoposide IV over 2 hours on days 1 and 2. Patients who are randomized to receive PSC 833 during induction chemotherapy receive a loading dose of PSC 833 before beginning a 48-hour continuous infusion of PSC 833 concurrently with cytarabine/daunorubicin/etoposide postremission chemotherapy.

After completing postremission chemotherapy, patients are randomized to a no further treatment group or interleukin-2 (IL-2) immunotherapy. Treatment begins within 5 months of postremission chemotherapy. IL-2 immunotherapy consists of low-dose subcutaneous (SC) IL-2 on days 1-14, 19-28, 33-42, 47-56, 61-70, and 75-90 and high-dose bolus SC IL-2 on days 15-17, 29-31, 43-45, 57-59, and 71-73.

Patients are followed every 2 months for 2 years, every 6 months for 2 years, annually until the tenth year, and then at relapse.

ELIGIBILITY:
Inclusion Criteria:

* Unequivocal histologic diagnosis of AML, FAB classification (M0-M7), excluding M3 (acute promyelocytic leukemia); patients with a history of antecedent myelodysplasia remain eligible for treatment on this trial
* No prior treatment for acute leukemia or myelodysplasia with four permissible exceptions:

  * Emergency leukapheresis;
  * Emergency treatment for hyperleukocytosis with hyroxyurea;
  * Cranial RT for CNS leukostasis (one dose only);
  * Growth factor/cytokine support.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 1998-01; Primary Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | From second randomization to relapse or death, assessed up to 10 years
  Analyzed by intention to treat.
Overall survival | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Maria Baer, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States

REFERENCES:
- [Derived] Seffernick AE, Mrozek K, Nicolet D, Stone RM, Eisfeld AK, Byrd JC, Archer KJ. High-dimensional genomic feature selection with the ordered stereotype logit model. Brief Bioinform. 2022 Nov 19;23(6):bbac414. doi: 10.1093/bib/bbac414. PMID 36184192
- [Derived] Mims AS, Kohlschmidt J, Borate U, Blachly JS, Orwick S, Eisfeld AK, Papaioannou D, Nicolet D, Mromicronzek K, Stein E, Bhatnagar B, Stone RM, Kolitz JE, Wang ES, Powell BL, Burd A, Levine RL, Druker BJ, Bloomfield CD, Byrd JC. A precision medicine classification for treatment of acute myeloid leukemia in older patients. J Hematol Oncol. 2021 Jun 23;14(1):96. doi: 10.1186/s13045-021-01110-5. PMID 34162404
- [Derived] Walker CJ, Kohlschmidt J, Eisfeld AK, Mrozek K, Liyanarachchi S, Song C, Nicolet D, Blachly JS, Bill M, Papaioannou D, Oakes CC, Giacopelli B, Genutis LK, Maharry SE, Orwick S, Archer KJ, Powell BL, Kolitz JE, Uy GL, Wang ES, Carroll AJ, Stone RM, Byrd JC, de la Chapelle A, Bloomfield CD. Genetic Characterization and Prognostic Relevance of Acquired Uniparental Disomies in Cytogenetically Normal Acute Myeloid Leukemia. Clin Cancer Res. 2019 Nov 1;25(21):6524-6531. doi: 10.1158/1078-0432.CCR-19-0725. Epub 2019 Aug 2. PMID 31375516